CLINICAL TRIAL: NCT02037776
Title: Double-blind Trial With Rikkunshito Versus Placebo on Efficacy and Safety in Patients With Functional Dyspepsia: Multi-center Study (DREAM Study)
Brief Title: The Efficacy and Safety Study of Rikkunshito in Patients With Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka City University (Other)
Responsible Party: Principal Investigator, Kazunari Tominaga, M.D., Ph.D., Osaka Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tj43-p2-t1
Record Dates: First submitted 2014-01-09; First posted 2014-01-16 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Functional Dyspepsia
Keywords: Rikkunshito; Double blind; Functional dyspepsia (FD)
MeSH Terms: interventions — liu-jun-zi-tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rikkunshito Placebo (Placebo Comparator)
  Interventions: Drug: Rikkunshito placebo
- Rikkunshito (Active Comparator)
  Interventions: Drug: Rikkunshito

INTERVENTIONS:
Drug: Rikkunshito — - Oral administration of rikkunshito (2.5 g t.i.d) before meals for 8 weeks
  Other Names: Tsumura Rikkunshito
  Arms: Rikkunshito
Drug: Rikkunshito placebo — - Oral administration of rikkunshito placebo (2.5 g t.i.d) before meals for 8 weeks
  Arms: Rikkunshito Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Rikkunshito compared to placebo in Japanese subjects with Functional Dyspepsia (FD).

ELIGIBILITY:
Inclusion Criteria:

* -Patients diagnosed with FD according to the ROME III criteria i) Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to obtaining informed consent ii) Have not received upper endoscopy within the last 6 months prior to enrollment and do not have evidence of structural/organic disease iii) Must have one or more of the following symptoms:

  1. Bothersome postprandial fullness
  2. Early satiation
  3. Epigastric pain
  4. Epigastric burning
* At least one of the FD-related symptoms on the Global Overall Symptom (GOS) scale (bothersome postprandial fullness, early satiation, epigastric pain, epigastric burning) is ≥4, whereas heartburn is ≤3.
* Total score of depression-related symptoms on Hospital Anxiety and Depression Score (HAD) is ≤10.
* Type of visit: Outpatient
* Provides voluntary informed consent after receiving adequate explanation and demonstrates thorough understanding of the nature of the study.

Exclusion Criteria:

* Confirmed ulcer (excluding scars) or malignant tumor in the upper GI
* Suspected organic lesions in the hepato-biliary-pancreatic regions such as cholelithiasis, hepatitis, pancreatitis
* History of upper GI resection
* Serious complications (liver, kidney, heart, or blood disease or metabolic disease)
* Less than a year since testing positive for H. pylori or have undergone a successful eradication therapy
* Use of prohibited medications
* Neuropsychiatric disorders
* Use of or planned use of any investigational drugs
* Unable to take drugs orally
* History of allergic reactions to Kampo medicines
* Pregnant or lactating women or those who are planning to conceive during the study period
* Deemed ineligible by principal investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuo Arakawa, Study Director — Osaka City University Graduate School of Medicine
Locations (1):
- Osaka City University Graduate School of Medicine, Abeno-ku, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rikkunshito Placebo | Rikkunshito
Started | 61 | 64
Completed | 56 | 60
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rikkunshito Placebo | Rikkunshito | Total
Number analyzed (Participants) | 61 | 64 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 53 | 102
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 50.4 (13.7) | 50.4 (14.9) | 50.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 42 | 89
  Male | 14 | 22 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 61 | 64 | 125
Subtype of functional dyspepsia (FD) [Count of Participants; unit: Participants] — The subtype of FD was diagnosed according to the Rome III Diagnostic Criteria for Functional Gastrointestinal Disorders. The Rome III criteria have divided functional dyspepsia into postprandial distress syndrome (PDS), characterized by postprandial fullness occurring after ordinary-sized meals at least several times per week and early satiation that prevents finishing a regular meal, at least several times per week, and epigastric pain syndrome (EPS), characterized by epigastric pain or burning of at least moderate severity at least once per week.
  Participants
    Postprandial distress syndrome (PDS) | 23 | 26 | 49
    Epigastric pain syndrome (EPS) | 18 | 24 | 42
    Both | 20 | 14 | 34
Duration of FD [Count of Participants; unit: Participants]
  ≥6 months to <1 year | 19 | 24 | 43
  ≥1 year | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Patient's Evaluation of Symptomatic Improvement by Overall Treatment Efficacy (OTE)
Description: Patient's Evaluation of Symptomatic Improvement by OTE is classified into the following 7 categories:
  1. Significantly improved
  2. Improved
  3. Slightly improved
  4. No change
  5. Slightly worse
  6. Worse
  7. Much worse
  The numbers of patients at the final evaluation (i.e, the latest evaluable time point of the all patients including discontinued patients) are shown by category.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rikkunshito Placebo | Rikkunshito
Number analyzed (Participants) | 61 | 64
Participants
  1=Significantly improved | 1 | 5
  2=Improved | 13 | 18
  3=Slightly improved | 25 | 26
  4=No change | 19 | 15
  5=Slightly worse | 3 | 0
  6=Worse | 0 | 0
  7=Much worse | 0 | 0
Statistical Analysis 1: Comparison: Rikkunshito Placebo vs Rikkunshito; Comparison between groups in Rikkunshito Placebo and Rikkunshito, based on the count of participants categorized in 1 (Significantly improved) through 7 (Much worse), using the Wilcoxon (Mann-Whitney); Test type: Superiority; p = 0.038, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Modified Frequency Scale for the Symptoms of Gastroesophageal Reflux Disease (GERD) (Modified FSSG)
Description: The modified FSSG questionnaire is composed of 7 questions regarding GERD symptoms (Questions 1-7, scored from 0 to 4) ranging between 0-28, lower value represents a better outcome, and 7 questions regarding dyspeptic symptoms (Questions 8-14, each question scored from 0 to 4) ranging between 0-28, lower value represents a better outcome, and a total scores, ranging from 0 to 56, lower value represents a better outcome of the all questions (Questions 1-14). Each question was assigned a score based on the frequency of symptoms.
  The point scores of modified FSSG are calculated from changes from baseline in each score for all symptoms (sum of point scores from Questions 1-14), GERD symptoms, and dyspeptic symptoms at final evaluation.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rikkunshito Placebo | Rikkunshito
Number analyzed (Participants) | 61 | 63
units on a scale
  All symptoms | -4.99 (5.92) | -7.18 (6.94)
  GERD symptoms | -1.69 (2.93) | -2.62 (4.07)
  Dyspeptic symptoms | -3.29 (4.25) | -4.58 (4.02)
Statistical Analysis 1: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in all symptoms of modified FSSG; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in GERD symptoms of modified FSSG; Test type: Superiority; p = 0.089, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in dyspeptic symptoms of modified FSSG; Test type: Superiority; p = 0.148, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM)
Description: PAGI-SYM questionnaire is composed of the following 6 categories that consisted of Questions 1 to 20 (each question composed of 6 subscales, i.e., point scores from 0 to 5, lower value represents a better outcome). Subscale scores are calculated by averaging across items in each category. A total score (lower value represents a better outcome, ranging from 0 to 5) is calculated as the mean of the subscale scores.
  Heartburn/Regurgitation, Nausea/Vomiting, Postprandial Fullness/Early satiety, Bloating, Upper Abdominal Pain, and Lower Abdominal Pain
  The point scores of PAGI-SYM are calculated from changes from baseline in total score and each category score at final evaluation.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rikkunshito Placebo | Rikkunshito
Number analyzed (Participants) | 61 | 63
units on a scale
  Total | -0.30 (0.43) | -0.47 (0.61)
  Heartburn/Regurgitation | -0.23 (0.48) | -0.25 (0.63)
  Nausea/Vomiting | -0.15 (0.75) | -0.33 (0.94)
  Postprandial Fullness/Early satiety | -0.36 (0.74) | -0.82 (0.98)
  Bloating | -0.20 (0.78) | -0.56 (1.00)
  Upper Abdominal Pain | -0.56 (1.20) | -0.76 (1.19)
  Lower Abdominal Pain | -0.31 (1.03) | -0.13 (0.90)
Statistical Analysis 1: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in total score of PAGI-SYM; Test type: Superiority; p = 0.051, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in Heartburn/Regurgitation of PAGI-SYM; Test type: Superiority; p = 0.947, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in Nausea/Vomiting of PAGI-SYM; Test type: Superiority; p = 0.157, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in Postprandial Fullness/Early satiety of PAGI-SYM; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in Bloating of PAGI-SYM; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in Upper Abdominal Pain of PAGI-SYM; Test type: Superiority; p = 0.245, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in Lower Abdominal Pain of PAGI-SYM; Test type: Superiority; p = 0.387, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in Global Overall Symptom (GOS)
Description: The GOS scale are calculated by a total score of a 7-point Likert scale ranging from 1 = no problem to 7 = a very severe problem over 8 questions. The point scores of GOS are calculated from changes from baseline at final evaluation.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rikkunshito Placebo | Rikkunshito
Number analyzed (Participants) | 61 | 64
units on a scale | -4.03 (5.08) | -6.39 (5.22)
Statistical Analysis 1: Comparison: Rikkunshito Placebo vs Rikkunshito; Test type: Superiority; p = 0.034, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Short-form Health Survey-8 (SF-8)
Description: The SF-8 scores comprised of Physical component summary (PCS) scores (ranging between 5.32-70.69, higher value represents a better outcome) and Mental component summary (MCS) scores (ranging between 10.11-74.51, higher value represents a better outcome), and a total scores of PCS and MCS using a formula specified in SF-8 Scoring Algorithm.
  The point scores of SF-8 are calculated from changes from baseline in PCS and MCS at final evaluation.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rikkunshito Placebo | Rikkunshito
Number analyzed (Participants) | 61 | 63
units on a scale
  PCS | 2.68 (5.84) | 3.87 (7.61)
  MCS | 0.24 (7.72) | 1.81 (6.58)
Statistical Analysis 1: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in PCS of SF-8; Test type: Superiority; p = 0.270, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in MCS of SF-8; Test type: Superiority; p = 0.342, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HAD)
Description: The HAD is a 14-item scale with 2 subscales of depression (Question 1, 3, 5, 7, 9, 11, and 13) and anxiety (Question 2, 4, 6, 8, 10, 12, and 14). Each item on the questionnaire is scored from 0 to 3 (ranging from 0 to 21, lower value represents a better outcome).
  The point scores of HAD are calculated from changes from baseline in overall (sum of scores for depression and anxiety, i.e., total point score ranging from 0 to 42, lower value represents a better outcome), depression, and anxiety at final evaluation.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rikkunshito Placebo | Rikkunshito
Number analyzed (Participants) | 61 | 64
score
  Overall | -0.34 (4.39) | -2.11 (5.05)
  Depression | -0.05 (2.85) | -0.92 (2.61)
  Anxiety | -0.30 (2.26) | -1.19 (3.03)
Statistical Analysis 1: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in overall point score of HAD; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in depression point score of HAD; Test type: Superiority; p = 0.084, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Rikkunshito Placebo vs Rikkunshito; Change from baseline in anxiety point score of HAD; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Rikkunshito Placebo | Rikkunshito
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 2/63 | 0/65
Other Adverse Events (participants affected / at risk) | 5/63 | 7/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rikkunshito Placebo (N=63) | Rikkunshito (N=65)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rikkunshito Placebo (N=63) | Rikkunshito (N=65)
Gingivitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fractures (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.